CLINICAL TRIAL: NCT00172406
Title: The Relation Between Serum Level of Amioterminal Propeptide of Type I Procollagen and Diastolic Dysfunction in Hypertensive Patients Without Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361700202
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
In the present study, we assessed the relation between diastolic dysfunction and myocardial fibrosis in hypertensive patients without diabetes mellitus. A total of 20 medically treated ambulatory non-diabetic hypertensive patients with normal left ventricular (LV) systolic function were enrolled into this study. Myocardial fibrosis was evaluated by serum concentrations of amino-terminal propeptides of type I and III procollagen (PINP and PIIINP). All patients underwent examinations of diastolic function by echocardiography and technetium-99m (99mTc) radionuclide ventriculography. There were 8 patients with PINP ≦53 μg/l (group 1) and 12 patients with PINP >53 μg/l (group 2). Patients in group 2 had significantly lower LV peak filling rate (PFR; 3.2 ± 0.3 vs. 2.5 ± 0.2 end-diastolic volume/s) and shorter time to PFR ( 257 ± 41 vs. 174 ± 22 ms). Besides, the group 2 patients also had lower right ventricle PFR (1.9 ± 0.2 vs. 1.5 ± 0.1 end-diastolic volume/s) and shorter time to PFR ( 221 ± 29 vs. 154 ± 29 ms). Echocardiographic parameters for LV diastolic dysfunction (E/A ratio of mitral flow, deceleration time of E flow, velocities of pulmonary venous flow [retrograde A wave, systolic /diastolic velocity ratio], isovolumetric relaxation time, Tei index) were all comparable between two groups. In multiple regression analysis, LV time to peak filling rate was the only parameter that independently predicted serum PINP level (p<0.05). In conclusion, elevated serum PINP level reflected LV diastolic dysfunction in hypertensive patients without diabetes.

ELIGIBILITY:
Inclusion Criteria:

* We enrolled 20 medically treated ambulatory, non-diabetic, hypertensive patients in this study.

Exclusion Criteria:

* Patients with abnormal liver functions, leukocytosis, elevated serum levels of C-reactive protein, systolic dysfunction (LV ejection fraction <50%) and LV hypertrophy due to etiologies other than hypertension were excluded from this study.

Min Age: 0 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Lwun Ho, MD, PhD, Principal Investigator — National Taiwan University Hospital